CLINICAL TRIAL: NCT03481686
Title: SelfEPO - Therapeutic Education of Chronic Renal or Renal Transplant Patient in the Management of EPO Injections
Brief Title: Therapeutic Education of Chronic Renal or Renal Transplant Patient in the Management of EPO Injections
Acronym: SELFEPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC16_9864_SELFEPO; 2017-A00295-48 (Other: N° ID - RCB)
Record Dates: First submitted 2018-03-19; First posted 2018-03-29 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Renal Insufficiency, Chronic; Organ Graft
Keywords: Erythropoiesis; stimulating; agents; therapeutic; education; program
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with injections of ESA (Experimental): Patients with injections of ESA
  Interventions: Device: Patients with injections of ESA

INTERVENTIONS:
Device: Patients with injections of ESA — Patients will perform ASE injections themselves or by their spouses

SUMMARY:
In chronic kidney disease, ESAs (Erythropoiesis-stimulating agents) are used to treat anemia. This anemia is due to decreased renal production of erythropoietin (EPO), a hormone that stimulates the production of red blood cells in the bone marrow. Treatment of anemia increases survival, decreases morbidity and improves quality of life and exercise tolerance.

Self-administration of ASE has been encouraged for many years, notably with pens for injection, but only few patients are educated in the injection technique.

The investigators therefore wish to lead a study in the Nephrology department of Rennes University Hospital to educate the patient, or his or her spouse, on ESA injections during hospitalization, in order to empower the patient in his care, and with the second aim of reducing the costs of chronic renal insufficiency.

DETAILED DESCRIPTION:
Erythropoiesis-stimulating agents (ESAs) are numerous and prescribed, depending on the molecule, once a week to once a month. They have improved the management of pre-dialysis patients, increased their hemoglobin and decreased transfusion needs, improving their morbidity and mortality and quality of life.

They are administered in pre-dialysis or post-renal transplantation most often by subcutaneous injection, which can be done by the patient himself, a member of his family or a nurse. Self-administration of ASE has been encouraged for many years, notably with pens for injection, but only few pilot studies show the feasibility of these auto-injections of ASE and patient satisfaction.

In 2012, the investigators conducted a practice study whose main objective was to have a picture of ESA injection practices for pre-dialysis patients. It is an observational, epidemiological, prospective and multicentric study, carried out by a questionnaire completed by the nephrologist during a consultation.

At the end of a 6-month collection period, 143 records were collected. All the patients questioned were followed for chronic renal insufficiency, not yet dialysed and not transplanted.

The majority of patients enrolled in this study were in the maintenance phase for ASE prescription (86% versus 14% in the correction phase), the mean age was 66.4 +/- 16.9 years. In 70.2% of cases the injection is done by a nurse, compared to 24.8% of injections made by the patient himself and 4.9% by his spouse. For 86.7%, the injection was done at home, and for 60% without other associated care. The nurse therefore came only for the injection of ASE. Not surprisingly, at an equal ASE cost, the resort to a nurse is significantly more expensive.

ELIGIBILITY:
Inclusion Criteria:

* Patients monitored for chronic renal failure, or for renal transplantation regardless of clearance level;
* Patients whose disease requires regular injections of ESA (before hospitalization or since hospitalization);
* Patients who did not realize their injection themselves before hospitalization;
* Patients hospitalized in the nephrology department at Rennes university hospital ;
* Obtaining free, informed and written consent;
* Affiliation to social security.

Exclusion Criteria:

* Major incapable persons and persons deprived of their liberty;
* Dialysis patients or for whom dialysis is envisaged within 3 months;
* Pregnant or nursing mothers;
* Patients who are already performing their ASE injections alone;
* Simultaneous participation in another research protocol involving the human person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Number of patients performing all their injections themselves and / or their spouse | 6 months

SECONDARY OUTCOMES:
Number of patients performing all their injections themselves | 1 month
Number of patients performing all their injections themselves | 3 months
Percentage of injections performed by the nurse vs by themselves and / or their spouse before empowerment | 6 months
Number of patients who performed all their injections by their spouse | 6 months
Number of injections performed on the number of prescribed injections | 6 months
  Treatment compliance
Injection site pain | 6 months
  pain assessment with a visual analog scale (0 = no pain, 10 = maximum pain)
Side effects of ESA injection | 6 months
Number of patients stopping self-injections | 6 months
Reason for stopping self-injections | 6 months
  evaluation of reason for stopping self-injections with a questionnaire
Number of patients refusing therapeutic education | 6 months
Reason for refusing therapeutic education | 6 months
  evaluation of reason for refusing therapeutic education with a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Cécile VIGNEAU, Principal Investigator — CHU Rennes; Hugoline BOULAY, Study Chair — CHU Rennes
Locations (1):
- CHU de Rennes, Rennes, France